CLINICAL TRIAL: NCT02874612
Title: Young Adults With Type 1 Diabetes: Psychosocial Influences in Heath Outcomes for Young Adults Transitioning to Adult Care Project
Brief Title: Psychosocial Functioning in Young Adults With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Baylor University (Other); Children's National Research Institute (Other); Texas A&M University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-1575
Record Dates: First submitted 2016-06-29; First posted 2016-08-22 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Young Adults; Psychosocial Functioning
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young Adults with Type 1 Diabetes Mellitus: All YA (ages 18-24) who are seen in the Cincinnati Children's Hospital Medical Center Diabetes Clinic and have recently (< 4 months) completed the Transition Readiness assessment tool as part of their standard clinical care is eligible for the study.
  Interventions: Other: Psychosocial Survey Questionnaires

INTERVENTIONS:
Other: Psychosocial Survey Questionnaires — Young adults with Type 1 Diabetes Mellitus will be invited to participate in a observational study in which they complete psychosocial measures immediately after completing a readiness transition survey and then again 1 year later.

SUMMARY:
Background: The often studied psychosocial correlates that relate to health outcomes in adolescents with Type 1 Diabetes (T1D) are factors such as self-efficacy, depression, distress, quality of life, and adherence. These psychosocial factors are not well-studied within a young adult (YA) population and the parents of YAs during the transition planning phase. Impact: This study aids program development for pre-transfer educational interventions to ensure more successful post-transfer health outcomes from both a patient and parent perspective. Methods: This longitudinal study is designed to characterize the psychosocial factors relevant for a population of YA with T1D. Data analyses of these psychosocial and transition readiness variables allow for understanding of prospective health outcomes for young adults with T1D during the transition process. Implications/Future Directions: From a clinical perspective, the outcomes of this feasibility study will be two-fold: (1) establish which of the clinical measures used in the study are related to meaningful health outcomes in this young adult population in order to determine future standardized assessments in the Diabetes Center and (2) determine which psychosocial constructs are relevant to health outcomes to then more fully develop the Diabetes Center's transition program interventions to improve functioning clinic-wide (e.g., group day sessions). Finally, it would be attractive to various National Institutes of Diabetes and Digestive and Kidney Disorder (NIDDK) grant mechanisms to identify the relevant psychosocial measures that assess the psychosocial functioning of YA with diabetes after they transfer to adult care.

DETAILED DESCRIPTION:
The purpose of this study is to assess how psychosocial functioning and transition readiness (health knowledge and self-reported health-related skills) of young adults (aged 18-24) with Type 1 Diabetes (T1D) and their parents impact health outcomes before they transition to adult diabetes care. Transition of health care from pediatric to adult care systems is a complex process and is often a challenge for young adults. These transition barriers lead to gaps in healthcare, worsening of glycemic control, and increased hospitalizations/emergency room utilization. Initial program development efforts to prepare young adults for transition were developed at Cincinnati Children's Hospital Medical Center (CCHMC) based on best practice recommendations in the literature. The psychosocial correlates of health outcomes in this population are not well studied, though. Nor is it known whether these diabetes education interventions impact transition to adult care over time. The investigators will study how psychosocial factors (e.g., self-efficacy, depression, distress, quality of life, adherence, and risky behaviors) impact health outcomes (e.g., glycemic control) over a one year period, within the context of the current diabetes education transition program at Cincinnati Children's Hospital Medical Center (CCHMC) for young adults with T1D and their parents.

ELIGIBILITY:
Inclusion Criteria:

* Young Adults ages 18-24
* Current patients of the Cincinnati Children's Hospital Medical Center (CCHMC) Diabetes Clinic
* Recently (< 4 months) completed the Readiness Assessment tool
* Planning to continue to receive diabetes services at CCHMC (i.e., not imminently being transferring their diabetes care to an adult provider) for the next 12 months.

Exclusion Criteria:

* Co-existing diagnosis of mental retardation or pervasive developmental disorder
* Not fluent in the English language.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All YA (ages 18-24) who are seen in the CCHMC Diabetes Clinic and have recently (< 4 months) completed the READdY assessment tool as part of their standard clinical care is eligible for the study. In addition, the YA will need to be planning to stay at CCHMC (i.e., not imminently being transferring their diabetes care to an adult provider) for the next 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2015-08; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Evidence of a correlation between negative diabetes health outcomes and psychosocial functioning over a 1 year period | 1 year
  Establish if and how the baseline psychosocial and transition readiness constructs relate to long-term health outcomes for young adults with T1D, over a 1 year time frame, which will guide future education interventions and anticipatory guidance for young adults transitioning to adult diabetes care.

SECONDARY OUTCOMES:
Number of participants rating themselves as having diabetes resilience as assessed by the Diabetes Resilience Measure (DRMY-YA) measure | 1 year
  Collaborate with Drs. Hilliard and Monaghan on their validation of the Diabetes Resilience (DRMY-YA) measure within a young adult with T1D population.
Number of participating rating themselves as having diabetes quality of life as assessed by the PedsQL Diabetes 3.2 measure | 1 year
  Collaborate with Dr. Varni on the validation of the PedsQL Diabetes 3.2 measure within a young adult with T1D population

CONTACTS AND LOCATIONS:
Overall Officials: Jessica C Kichler, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de-identified data will be shared with the collaborating institutions and is outlined in the consenting process.